CLINICAL TRIAL: NCT01635569
Title: Clinical Outcomes Following Group-based Family Cognitive-Behaviour Therapy in Pediatric Obsessive-Compulsive Disorder (OCD)
Brief Title: Clinical Outcomes in Pediatric Obsessive-Compulsive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Michael Smith Foundation for Health Research (Other)
Responsible Party: Principal Investigator, Evelyn Stewart, MD, Principle Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H12-01656
Record Dates: First submitted 2012-06-27; First posted 2012-07-09 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Obsessive-compulsive Disorder
Keywords: Obsessive-compulsive disorder; Pediatric; Group-based; Cognitive-behavioural therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OCD-affected subjects (Group 1) (Active Comparator): OCD-affected subjects will participate in 12 sessions of group therapy (as per GF-CBT protocol).
  Interventions: Behavioral: Group-based family cognitive-behavioural therapy
- OCD-affected subjects (Group 2) (Active Comparator): Waitlist affected-controls awaiting a treatment spot.
  Interventions: Other: Waitlist

INTERVENTIONS:
Behavioral: Group-based family cognitive-behavioural therapy — Baseline and post-12 sessions
  Arms: OCD-affected subjects (Group 1)
Other: Waitlist — Baseline and post-12 sessions
  Arms: OCD-affected subjects (Group 2)

SUMMARY:
Obsessive-Compulsive Disorder (OCD) is a common neuropsychiatric illness beginning in childhood. Effective OCD treatments include cognitive-behaviour therapy (CBT) and medications but access to treatment is difficult and does not systematically include parents. The investigators will evaluate clinical and neural effects of Group-based Family CBT (GF-CBT), via a case-control study including: Group 1 - OCD cases receiving GF-CBT (N=90); Group 2 - OCD waitlist cases (N=90). Effects will be measured between baseline and completion of 12 GF-CBT sessions: comparing OCD severity and functioning changes between Groups 1 and 2.

DETAILED DESCRIPTION:
Effective OCD treatment approaches in children and youth include cognitive-behaviour therapy (CBT) and serotonergic medications; however, the disorder is under-diagnosed and access to care is frequently delayed or difficult to obtain. Moreover, despite the important role of family accommodation as an outcome predictor, standard CBT does not systematically include parents and mechanisms of response are not fully understood. The investigators propose to address this challenge by evaluating a novel treatment approach called Group-based Family CBT (GF-CBT).

To determine clinical and neural effects of GF-CBT, we will perform a case-control study of two groups: Group 1 - OCD-affected youth receiving GF-CBT treatment (N=90); Group 2 - OCD-affected youth receiving no new treatment (waitlist controls; N=90).

The investigators will collect clinical outcome data related to OCD severity, individual and family functioning at four time points for Group 1 subjects and at two time points for Group 2 subjects. For Group 1 subjects, these time points include baseline, at midpoint, at the completion of 12 sessions, and at one-month follow-up (all time points are +/- one week). For Group 2 subjects, time points will be at baseline and after a time delay equivalent to completion of 12 GF-CBT sessions. Clinical measures will be used to compare changes between GF-CBT treatment and waitlist-control groups (Groups 1 versus 2).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 5-18 years old
* Ability of subject and parent to provide informed assent/consent
* English-speaking
* Current DSM IV-TR Axis I diagnosis of childhood-onset OCD; Moderate to severe OCD (CY-BOCS≥16/40)

Exclusion Criteria:

* Current diagnosis of bipolar disorder, psychosis, mental retardation or pervasive developmental disorder (e.g., autism), and current or past substance dependence/abuse

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2012-10-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Children's Yale Brown Obsessive-Compulsive Scale (CY-BOCS) | Baseline, midpoint, completion of 12 GF-CBT sessions, one-month follow-up
  CY-BOCS: gold-standard measure of OCD severity in pediatric OCD.

CONTACTS AND LOCATIONS:
Overall Officials: S. Evelyn Stewart, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada